CLINICAL TRIAL: NCT07267910
Title: Measuring Vestibular Organ Function With Weak Alternating-current Stimulation
Brief Title: Measuring Vestibular Organ Function With Weak Alternating Current Stimulation
Acronym: VESTI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalto University (Other)
Collaborators: Helsinki University Central Hospital (Other); Business Finland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VESTI
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Vestibular Disorder; Vestibular Schwannoma; Vestibular Neuritis
Keywords: Vestibular disorders; Otorhinolaryngologic Diseases; Electrical vestibular stimulation; transcranial electrical stimulation
MeSH Terms: conditions — Vestibular Diseases; Neuroma, Acoustic; Vestibular Neuronitis; Otorhinolaryngologic Diseases

STUDY DESIGN:
Intervention Model Description: All study participants will get the same interventions but in different randomized order. The order randomization is based on the balanced Latin square design such that each intervention type occurs equally often in each position in the order, so that any order effects are distributed evenly among the subjects.
Masking Description: All study participants will get the same interventions but in different randomized order. The investigator does know the possible types of intervention but not the order they will be applied in. Therefore at the time of applying the intervention neither the participant nor the investigator know which specific intervention is being applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EVS + measurement (Experimental): The study composes of multiple interventions (1-3 min electrical vestibular stimulation and response measurement). All study participants will get the same interventions but in different randomized order.
  Interventions: Device: Active transcranial electrical vestibular stimulation (Active EVS); Device: Sham transcranial electrical vestibular stimulation (Sham EVS); Device: Control measurement

INTERVENTIONS:
Device: Active transcranial electrical vestibular stimulation (Active EVS) — Active transcranial electrical vestibular stimulation (EVS) with alternating current (maximum peak current below 2 mA and stimulation frequency 2-20 Hz) applied for 1-3 minutes at a time and for under 20 minutes in total. EVS will be applied either bilaterally (ear to ear) or unilaterally (left ear to neck or right ear to neck). The participants movements during the stimulation are measured with a force plate and wearable acceleration sensors. The study uses multiple types of vestibular stimulation waveforms which are applied in a randomized sequence, such that neither the participant nor the investigator know the exact stimulation type at the time of the measurement.
Device: Sham transcranial electrical vestibular stimulation (Sham EVS) — Sham (no current) transcranial electrical vestibular stimulation applied for 1-3 minutes. The participant's movements during the supposed stimulation are measured with a force plate and wearable acceleration sensors. Neither the participant nor the investigator know at what point of the intervention sequence the sham stimulation is applied.
Device: Control measurement — The participant's movements are measured with a force plate and wearable acceleration sensors for the same time duration (1-3 min) and following the same protocols as in other interventions, but both the participant and the investigator know that no stimulation is being applied. The control measurement will always be completed before all other interventions and is not part of the randomized intervention sequence.

SUMMARY:
The goal of this clinical trial is to preliminarily evaluate the use of electrical stimulation in diagnosing disorders with the vestibular system. The main questions it aims to answer are:

* Can electrical vestibular stimulation combined with movement measurement be used to diagnose disorders of the vestibular system?
* Can electrical stimulation provide treatment or rehabilitation opportunities for patients suffering from disorders of the vestibular system?

DETAILED DESCRIPTION:
The participants will each attend one experimental session consisting of multiple short (1-3 min) measurement trials. During a trial the participant's vestibular system is stimulated with a transcranial electrical stimulator device and their movements are recorded with a force plate and acceleration sensors.

The goal of the study is to collect and analyse data from 30 research participants with diagnosed vestibular disorders.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* One of the following: clinically diagnosed vestibular schwannoma, vestibular neuritis, or simultaneous unilateral hearing loss and vestibular dysfunction.

Exclusion Criteria:

* History of epilepsy or seizures
* Past brain surgery
* Pacemaker, cochlear implant, or other implanted medical device
* Pregnancy
* Skin problems or damaged skin at the site of the stimulation (scalp and neck)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Changes in the frequency content of the movement response signals | From study appointment to the analysis of the results (up to 12 months)
  Changes of the power in a frequency band of 0-20 Hz in the measured movement response signals during active electrical vestibular stimulation (EVS). The measured movement response signals are force plate Center of Pressure (CoP) and 3-axis acceleration data from wearable acceleration sensors.

SECONDARY OUTCOMES:
Latency of the EVS response | From study appointment to the analysis of the results (up to 12 months)
  Latency of the EVS-induced movement response measured as the time delay between the stimulation and the measured movement.
Highest frequency of the EVS-induced response | From study appointment to the analysis of the results (up to 12 months)
  Highest frequency at which EVS induces a response determined via spectral analysis of the movement data

CONTACTS AND LOCATIONS:
Overall Officials: Ilkka Laakso, D.Sc. (Tech), Principal Investigator — Aalto University; Topi Jutila, MD, PhD, Principal Investigator — HUS Helsinki University Hospital
Locations (1):
- Dept. of Otorhinolaryngology, HUS Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No